CLINICAL TRIAL: NCT06394180
Title: PeRforation EVents During ENdovascular Therapy for Acute Ischemic Stroke (PREVENT) - Registry
Brief Title: PeRforation EVents During ENdovascular Therapy for Acute Ischemic Stroke
Acronym: PREVENT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 0000-00000; th23Psychogios2
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Periprocedural Vessel Perforation; Acute Ischemic Stroke
Keywords: Registry; Thrombectomy Complications; Endovascular Hemostatic Therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perforation during thrombectomy: The target cohort includes 500 patients where vessel perforation occured during Thrombectomy.
- No perforation during thrombectomy: The comparison cohort includes 500 patients, matched to the target cohort, where vessel perforation did not occur during Thrombectomy.

SUMMARY:
A large, worldwide study called PREVENT is looking at a complication that can happen during a stroke treatment called thrombectomy. This complication is a perforation of a blood vessel. The investigators aim to:

1. Find what factors make this perforation more likely.
2. Understand why the perforation happens by looking closely at images taken during the procedure.
3. Create a simple way to classify these perforations to help doctors decide how to treat them right away.
4. Improve the emergent treatment of vessel perforation to stop the bleeding rapidly.
5. Provide data to guide decision whether thrombectomy should be continued or aborted after the event of vessel perforation.
6. Develop a safer way to perform thrombectomy.

Investigators will compare the results collected for patients where perforation happened with those where perforation did not happen.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and the leading cause of disability, both worldwide and in Europe. Endovascular treatment (ENT), also called thrombectomy, is a minimally invasive procedure in which the occlusion of the brain-supplying artery, which is the cause of the stroke, is recanalized by removing the obstructing blood clot using endovascular methods, i.e. via access through the vessels, and thus restoring blood flow in the affected vessel and re-establishing brain perfusion. In 2015, five randomized controlled trials showed an overwhelming benefit of thrombectomy in patients with acute ischemic stroke with large vessel occlusion of the anterior circulation with a number needed to treat as low as 2.6. Since then, the indications for thrombectomy have been expanding continuously, including patients with posterior circulation occlusions, selected patients presenting late after symptom onset and patients with large infarcts. In addition, patients with distal vessel occlusions are increasingly being considered for thrombectomy.

Despite the effectiveness of thrombectomy, the procedure has a relevant risk of periprocedural complications. In 1-2% of patients who undergo thrombectomy, a periprocedural intracranial vessel perforation occurs with subsequent arterial intracranial bleeding. This complication typically represents a major turning point and is associated with severe permanent sequelae and a mortality of approximately 50%. Given the rapidly increasing frequency of thrombectomies, an increase in the incidence of periprocedural perforations is to be expected. The available data on vascular perforations during thrombectomy are limited. It is unknown why a minority of patients experience this complication while the majority are spared. Likewise, the exact pathophysiological process that leads to vessel wall damage is not understood. There is also uncertainty as to whether extravasation in the event of vessel perforation should be treated endovascularly with intention to stop the bleeding, e.g. via temporary vessel occlusion using a balloon catheter or permanent vascular occlusion using coils or liquid embolization. In addition, there is hardly any data on whether thrombectomy attempts should continue after a perforation has occurred or whether the procedure should be aborted. Due to the low frequency of this complication, randomized prospective trials will most likely not be feasible.

In an international retrospective cohort study with 25 participating centers, the investigators were able to evaluate data from over 25,000 thrombectomies. In this cohort, 335 vessel perforations were reported. About half of the affected patients died within the first 3 months after perforation. The remaining patients experienced a clinical course that was, on average, worse than that of stroke patients without perforation in large registries. This research represents the largest cohort of patients with perforation during thrombectomy to date. It shows that although perforations are rare complications, they have enormous relevance for the affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of thrombectomy
* Acute ischemic stroke with occlusion of one or several intracranial arteries and subsequent thrombectomy.
* Target cohort: Occurrence of intracranial perforation during thrombectomy with evidence of contrast extravasation in at least one diagnostic angiography series.
* Comparison cohort: No perforation during thrombectomy. Every patient in the comparison group is matched to one patient in the target population. Matching will be carried out with respect to age, gender, participating center and location of the vascular occlusion.

Exclusion Criteria:

* Presence of a documented rejection
* Presence of both ischemic stroke and intracranial hemorrhage on pre-interventional imaging.
* Patients with intracranial dissection without active contrast extravasation.
* Patients with rupture of a pre-existing intracranial aneurysm during thrombectomy.
* Patients with contrast medium extravasation into a venous space instead of free contrast medium extravasation, e.g. the cavernous sinus with consecutive development of a carotid-cavernous fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without vessel perforation perforation during thrombectomy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days
  The mRS is a measure of patient global disability. The scale is coded from 0 (no symptoms at all) through 5 (severe disability) and 6 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Schulze-Zachau, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schulze-Zachau V, Rommers N, Muenger H, Singh GK, Katan M, Balmer L, Psychogios S, Brehm A, Fischer U, Psychogios MN. PREVENT: Towards the prevention of intracranial vessel perforations during mechanical thrombectomy - protocol for a multicenter registry study. Front Neurol. 2026 Jan 23;16:1680379. doi: 10.3389/fneur.2025.1680379. eCollection 2025. PMID 41659979